CLINICAL TRIAL: NCT03325855
Title: Fecal Microbiota Transplant National Registry
Acronym: FMT
Status: Recruiting | Type: Observational
Sponsor: American Gastroenterological Association (Other)
Collaborators: OpenBiome (Industry); University of California, San Diego (Other); University of Pennsylvania (Other); University of Minnesota (Other); Loyola University Chicago (Other); Commure, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: AmericanGA
Record Dates: First submitted 2017-10-17; First posted 2017-10-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Fecal Microbiota Transplantation; Clostridium Difficile Infection; Gut Microbiome
Keywords: FMT; CDI; Fecal Matter Transplant
MeSH Terms: conditions — Clostridium Infections | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None - Observational — None - Observational
  Other Names: Observational

SUMMARY:
A national data registry of patients receiving fecal microbiota transplantation (FMT) or other gut-related-microbiota products designed to prospectively assess short and long-term safety and effectiveness

DETAILED DESCRIPTION:
This registry will prospectively enroll 4,000 patients who undergo FMT at 75 sites throughout North America. Information on FMT methodology employed (e.g., screening of donor and recipient, preparation, FMT delivery) will be collected from each site. The indication for FMT as well as baseline information on recipient will also be collected. Following FMT, patients will be followed at regular intervals up to 10 years post FMT. This will include follow-up information from the patient's healthcare provider at 1 month, 6 months, 1 year, and 2 years after FMT as well as direct communication with patients at least annually up to 10 years after FMT. Follow-up information collected will be designed to assess potential short-term and long-term safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Recipient Inclusion Criteria

  * Ability to give informed consent
  * Receiving FMT or other gut-related microbiota product within 90 days after providing consent
  * Access to internet and/or telephone
* Donor Inclusion

  * Ability to give informed consent
  * Providing stool sample for FMT

Exclusion Criteria:

* Incarceration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving FMT or other gut-related-microbiota products and the donors providing specimens for the enrolled patients' FMT. Patients will be enrolled regardless of race, gender, ethnicity, or age.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related Adverse Events | over 10 Years
  Adverse events to be monitored include surgeries, infection, hospitalization, other life-threatening events, death and newly diagnosed diseases.
Disease Re-occurrence Following FMT | over 10 Years
  Assess effectiveness of FMT by monitoring disease re-occurrence post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Wu, MD, Principal Investigator — Co-Director, PennCHOP Microbiome Program; Colleen Kelly, MD, Principal Investigator — Brigham and Women's Hospital; Loren Laine, MD, Principal Investigator — Yale University
Locations (53):
- United States (52):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, Los Angeles, California
  - Stanford University, Redwood City, California
  - Sutter Roseville Medical Center, Roseville, California
  - University of California San Francisco, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - Yale New Haven Hospital, Hamden, Connecticut
  - MedStar Georgetown University Hospital, Georgetown, District of Columbia
  - Best Quality Research, Inc., Hialeah, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - GI Pros, Naples, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - University of Chicago School of Medicine, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Loyola University of Chicago/ Loyola University Medical Center, Maywood, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Ochsner, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - American Gastroenterological Association, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Memorial Health, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health Hospital, Detroit, Michigan
  - Mayo Clinic - Division of Pediatric Gastroenterology, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Valley Hospital and Medical Center, Las Vegas, Nevada
  - Atlantic Health System, Morristown, New Jersey
  - Rutgers, New Brunswick, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Concorde Medical Group, New York, New York
  - New York University School of Medicine, New York, New York
  - Weill Cornell Medicine - Pediatric, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Gastroenterology Group of Rochester, LLP, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - Brown University Women's Medicine and Collaborative, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - Baylor Research Institute - Scott & White Medical Center, Temple, Texas
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Alberta, Edmonton, Alberta, Canada

DOCUMENTS (1):
  • Study Protocol (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03325855/Prot_000.pdf